CLINICAL TRIAL: NCT07360431
Title: Preoperative Granisetron in Combination With Dexamethasone or Metoclopramide for Prevention of Postoperative Nausea and Vomiting in Female Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Granisetron Combined With Dexamethasone or Metoclopramide for PONV Prevention After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amir Mohamed Abd El Halim Mokhimar, Anesthesiogy Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GRAN-PONV-LC
Record Dates: First submitted 2025-12-24; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-group clinical trial evaluating the preventive effect of granisetron plus dexamethasone versus granisetron plus metoclopramide on the prevention of postoperative nausea and vomiting in female patients undergoing laparoscopic cholecystectomy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design with identical preparation and administration of study medications to maintain blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Granisetron + Dexamethasone (Experimental): Patients will receive granisetron preoperatively, followed by dexamethasone administered after induction of anesthesia for prevention of postoperative nausea and vomiting.
  Interventions: Drug: Granisetron
- Granisetron + Metoclopramide (Experimental): Patients will receive granisetron preoperatively, followed by metoclopramide administered after induction of anesthesia for prevention of postoperative nausea and vomiting.
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Granisetron — Granisetron will be administered intravenously preoperatively for prevention of postoperative nausea and vomiting in female patients undergoing laparoscopic cholecystectomy.

SUMMARY:
Postoperative nausea and vomiting (PONV) remain common and distressing complications following laparoscopic cholecystectomy, particularly in female patients. This randomized interventional study aims to evaluate the effectiveness of preoperative granisetron when combined with either dexamethasone or metoclopramide in preventing PONV. The study compares the incidence and severity of nausea and vomiting, as well as the need for rescue antiemetic therapy, among female patients undergoing laparoscopic cholecystectomy under general anesthesia.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are among the most frequent complications after laparoscopic cholecystectomy and are associated with patient discomfort, delayed recovery, prolonged hospital stay, and decreased patient satisfaction. Female gender, laparoscopic surgery, and the use of general anesthesia are well-recognized risk factors for PONV.

Granisetron, a selective 5-hydroxytryptamine type 3 (5-HT3) receptor antagonist, has proven efficacy in the prevention of PONV. Combining granisetron with other antiemetic agents that have different mechanisms of action, such as dexamethasone or metoclopramide, may enhance its antiemetic effect through a multimodal approach.

This prospective randomized interventional study is designed to compare the efficacy of preoperative granisetron combined with dexamethasone versus granisetron combined with metoclopramide in preventing PONV in female patients undergoing laparoscopic cholecystectomy under general anesthesia. Eligible patients will be randomly allocated into two groups to receive either granisetron with dexamethasone or granisetron with metoclopramide prior to induction of anesthesia.

The primary outcome measure will be the incidence of postoperative nausea and vomiting within the first 24 hours after surgery. Secondary outcomes will include the severity of nausea, frequency of vomiting episodes, requirement for rescue antiemetic medications, and the occurrence of any adverse effects related to the study drugs.

The results of this study aim to identify the more effective granisetron-based combination for PONV prophylaxis in this high-risk population, potentially contributing to improved postoperative care and patient satisfaction following laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

- 1- Adult female. 2- (ASA I-II), aged 18-60 years. 3- Non smoker. 4- Scheduled for elective laparoscopic cholecystectomy under general anesthesia.

5- Use of intraoperative opioid analgesics.

Exclusion Criteria:

* 1- History of hypersensitivity to study drugs. 2- Chronic antiemetic. 3- Antidepressant use. 4- Gastrointestinal disease. 5- Pregnancy/lactation. 6- Severe hepatic/renal dysfunction

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study includes female participants only.
Enrollment: 102 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) | 0-24 hours postoperatively
  The incidence of postoperative nausea and vomiting (PONV) will be recorded and compared between the two study groups.

SECONDARY OUTCOMES:
Severity of postoperative nausea | 0-24 hours postoperatively
  Severity of nausea will be assessed using a visual analog scale (VAS) ranging from 0 to 10.
Number of vomiting or retching episodes | 0-24 hours postoperatively
  The total number of vomiting or retching episodes will be recorded for each patient.
Requirement for rescue antiemetic medication | 0-24 hours postoperatively
  The need for rescue antiemetic medication will be recorded during the postoperative period.
Patient satisfaction score | 0-24 hours postoperatively
  Patient satisfaction with postoperative nausea and vomiting management will be assessed using a satisfaction scoring system.
Incidence of adverse effects | 0-24 hours postoperatively
  The incidence of adverse effects including headache, dizziness, and extrapyramidal symptoms will be recorded.

IPD SHARING:
Plan to Share IPD: No